CLINICAL TRIAL: NCT04772794
Title: Immunological Effect of Intraoperative Fraction of Inspired Oxygen in Patients Undergoing Major Abdominal Cancer Surgery
Brief Title: Immunologic Effect of Fraction of Inspired Oxygen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, Associate Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 519
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Immune System
Keywords: fraction of inspired oxygen; hyperoxia; immune system
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyperoxygenation group (Active Comparator): Intraoperative administration of a mixture of 80% oxygen and 20% air
  Interventions: Other: fraction of inspired oxygen
- control group (Placebo Comparator): intraoperative administration of 30% oxygen and 70% air
  Interventions: Other: fraction of inspired oxygen

INTERVENTIONS:
Other: fraction of inspired oxygen — after induction of general anaesthesia, different fraction of inspired oxygen will be given to patient according to their group allocation

SUMMARY:
During anesthesia and surgery, oxygen is routinely administered to all patients. Inspired oxygen concentrations, however, vary between 30% - 100% and oxygen is often administered in a seemingly random manner.

DETAILED DESCRIPTION:
During anesthesia and surgery, oxygen is routinely administered to all patients. Inspired oxygen concentrations, however, vary between 30% - 100% and oxygen is often administered in a seemingly random manner.A striking conundrum is evident immediately when one review studies on the effects of oxygen on cytokines synthesis. Most investigators have found that hyperoxia enhances proinflammtory cytokines transcription and translations (11). In contrast, hyperparic oxygen has generally been shown to suppress stimulus induced porinflammtory cytokine production (12). Other studies have demonstrated that supplemental oxygen improves inflammatory and immune function (13), and it is not associated with clinically important side effect (14). We therefor undertook the current prospective randomized study to investigate whether perioperative supplemental oxygen (30% versus 80%) on pro and anti-inflammatory response in patients undergoing major abdominal cancer surgeries as our primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* candidates for abdominal cancer surgeries

Exclusion Criteria:

* Patients with chronic diseases, such as chronic obstructive pulmonary disease or pneumonia,
* body mass index (BMI) >35 kg/m2,
* severe malnutrition (albumin <3),
* leukopenia (white blood cell <4,000 g/dL),
* surgery within the previous 30 days and
* O2 saturation < 90%, as measured using a pulse oximeter

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
changes in serum level of interlukin 6 | before operation (0), 1st, 3rd, and 7th days postoperative
  serum level of interlukin 6 will be measured by ELISA technique
changes in serum level of interlukin 10 | before operation (0), 1st, 3rd, and 7th days postoperative
  serum level of interlukin 6 will be measured by ELISA technique

SECONDARY OUTCOMES:
changes in total WBCs count | before operation (0), 1st, 3rd, and 7th days postoperative
  measurement of total white blood cells count

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt